CLINICAL TRIAL: NCT01928004
Title: Implant-supported Mandibular Overdentures in Very Old Adults - a Randomized Controlled Trial
Brief Title: Mandibular Implants in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Frauke Müller, Professor and Chair, University of Geneva, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDGPA_02; ITI_458_2006 (Other Grant/Funding Number: International Team of Implantology ITI)
Record Dates: First submitted 2013-08-16; First posted 2013-08-23 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Edentulous Complete Denture Wearers
Keywords: edentulous; complete denture
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- implant placement (Experimental): insertion of 2 interforaminal mandibular implants and conversion of the lower complete denture to an implant-overdenture
  Interventions: Device: Implant placement
- denture reline (Active Comparator): conventional reline of mandibular complete denture
  Interventions: Procedure: Conventional reline

INTERVENTIONS:
Device: Implant placement — Participants received two Straumann Standard Implants® in the interforaminal region using the recommended surgical protocol. The implants were loaded using Locator® attachments after six to eight weeks healing time by transforming the existing lower denture to an IOD.
  Other Names: Straumann Standard Implants® (SLA surface, 8mm length, RN, 4.1mm diameter); Locator® attachments (Zest Anchors: Escondido, CA, USA)
  Arms: implant placement
Procedure: Conventional reline — conventional reline of the existing mandibular complete denture
  Arms: denture reline

SUMMARY:
The purpose of this study is to investigate denture satisfaction following the conversion of existing mandibular complete dentures to implant-overdentures (IOD) in very old edentulous patients who depend on help for activities of daily living (ADL) and evaluate secondary endpoints such as functional, structural, nutritional, cognitive and patient-centered outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* 75 years or older
* living institutionalized or receiving help for the ADL
* edentulous
* wearing complete dentures
* the lower denture had to cause discomfort to the degree that the patients were seeking treatment

Exclusion Criteria:

* severe clinical depression
* dementia
* poorly controlled diabetes
* immunosuppression
* treatment with bisphosphonates
* condition precluding the surgical intervention for implant placement

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-09; Primary Completion 2012-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Denture satisfaction | at 3, 12, 24 and 36 months
  VAS-scale score to evaluate the subjective satisfaction with the denture

SECONDARY OUTCOMES:
Change from Baseline in OHRQoL | at 3, 12, 24 adn 36 months
  OHIP-Edent questionnaire, 20 questions
Change from Baseline in cognitive function | at 12, 24 and 36 months
  Mini-Mental State Examination, to evaluate cognitive function (Folstein et al. 1975) Trail-making test A and B Verbal fluency test
Change from Baseline in Independence | at 12, 24 and 36 months
  IADL Instrumental Activities of Daily Living Scale (Lawton and Brody, 1969) MIF Measure of functional independence
Change from Baseline in MNA | at 3, 12, 24 and 36 months
  Mini-nutritional Assessement questionnaire (Guigoz 1994)
Change from Baseline in Blood markers | at 3, 12, 24 and 36 months
  Albumin, Folic acid, Vitamin B12 (VitB12), Hemoglobin (Hb), C-reactive protein (CRP)
Change from Baseline in BMI | at 12, 24 and 36 months
  Body Mass Index kg/m2
Change from Insertion in implant survival | at 3, 12, 24 and 36 months
  inserted implants in vivo
Change from Insertion in Pocket depth | at 3, 12, 24 and 36 months
  mesial and distal peri-implant probing depth
Change from Insertion in Plaque index | at 3, 12, 24 and 36 months
  Plaque index on implants (Silness & Loe 1963) Denture plaque index
Change from Insertion in peri-implant bone loss | at 3, 12, 24 and 36 months
  mesial and distal peri-implant bone loss, as evaluated on intraoral radiographs or OPTs
Change from Baseline in Chewing efficiency | at Intervention, 3, 12, 24 and 36 months
  two color mixing test with bi-colored chewing gum (Schimmel et al 2007)
Change from Baseline in Maximum bite force | at Intervention, 3, 12, 24 and 36 months
  unilateral maximal bite force measured with force gauge
Change from Baseline in Stimulated Saliva Flow Rate | at Intervention, 3, 12, 24 and 36 months
  whole saliva collected after chewing wax for 2 minutes on one side
Changes from Baseline in Masseter Muscle Thickness | at 3, 12, 24 and 36 months
  ultrasound measurements of the masseter muscle thickness in contracted and relaxed state

CONTACTS AND LOCATIONS:
Overall Officials: Frauke Müller, Prof. Dr. med. dent., Principal Investigator — University of Geneva
Locations (1):
- University of Geneva, Geneva, Switzerland

REFERENCES:
- [Result] Muller F, Duvernay E, Loup A, Vazquez L, Herrmann FR, Schimmel M. Implant-supported mandibular overdentures in very old adults: a randomized controlled trial. J Dent Res. 2013 Dec;92(12 Suppl):154S-60S. doi: 10.1177/0022034513509630. Epub 2013 Oct 24. PMID 24158342
- [Result] Maniewicz S, Duvernay E, Srinivasan M, Perneger T, Schimmel M, Muller F. Effect of implant-supported mandibular overdentures versus reline on masticatory performance and salivary flow rates in very old adults-A randomized clinical trial. Clin Oral Implants Res. 2019 Jan;30(1):59-67. doi: 10.1111/clr.13392. Epub 2018 Dec 30. PMID 30500094